CLINICAL TRIAL: NCT04340479
Title: The Use of Ultrasound in Establishing COVID-19 Infection as Part of a Trauma Evaluation
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0751
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: COVID; Trauma; Ultrasound
Keywords: COVID; Trauma; Ultrasound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Absent lung ultrasound findings of active COVID infection: Absence of bilateral, diffuse pleural line abnormalities, subpleural consolidations, white lung areas and thick, irregular vertical artifacts
  Interventions: Diagnostic Test: Ultrasound lung imaging as part of FAST+ evaluation
- Present lung ultrasound findings of active COVID infection: Presence of bilateral, diffuse pleural line abnormalities, subpleural consolidations, white lung areas and thick, irregular vertical artifacts
  Interventions: Diagnostic Test: Ultrasound lung imaging as part of FAST+ evaluation

INTERVENTIONS:
Diagnostic Test: Ultrasound lung imaging as part of FAST+ evaluation — FAST+ evaluations will expand on the traditional FAST exam to systematically survey bilateral lung fields. Traditional FAST evaluation will survey the perihepatic, perisplenic, pelvic, and pericardial areas. Representative images will be saved by the performing provider for further evaluation. Up to sixteen areas in total will be included in FAST+ evaluation:
  1. Anterior midclavicular right and left (apical, medial, basal)
  2. Posterior paraspinal right and left* (apical, medial, basal)
     *Posterior lung evaluation will be omitted if patients are at risk for further traumatic injury from repeated side rolling.
  3. Lateral axillary medial right and left (apical and basal)
  Specifically, we will document the presence or absence of bilateral, diffuse pleural line abnormalities, subpleural consolidations, white lung areas and thick, irregular vertical artifacts in these lung fields by ultrasound and will record these findings.

SUMMARY:
The current COVID-19 pandemic is providing healthcare organizations with considerable challenges and opportunities for rapid cycle improvement efforts, in diagnostic and patient management arenas. Healthcare providers are tasked with limiting the use of personal protective equipment while minimizing unnecessary exposures to the virus. Results from real-time PCR tests to detect active COVID-19 infections may not be available in a timely fashion during emergent trauma assessments. Since the start of the COVID-19 pandemic, a rapidly expanding body of literature has identified a pattern of imaged lung abnormalities with CT and ultrasound (US) characteristic of an active viral infection. US evaluation provides a reliable, portable, and reproducible way of evaluating acute patients in a real time setting. During initial trauma evaluations, patients may also receive adjunct imaging modalities like the Focused Assessment with Sonography in Trauma (FAST) exam designed to discover life threatening findings that may require urgent interventions. We therefore propose a study expanding on the current FAST adjunct evaluation in the trauma bay that may include lung parenchyma imaging at the initial assessment to help stratify patients into low or high-risk groups for active COVID-19 infections. We believe the use of point of care US in the initial assessment of the trauma patient may help identify potentially infected individuals and aid ED providers to best directing subsequent laboratory and imaging evaluations for these patients, while further directing the necessary protective measures for additional team members involved in the care of the injured patient.

DETAILED DESCRIPTION:
The current coronavirus disease 2019 (COVID-19) pandemic has created a unique situation for initial healthcare providers who strive to provide optimal medical care while minimizing personal exposure in acute scenarios. Although the morbidity and mortality for this disease is low for young healthy individuals, it presents a potentially serious threat to older healthcare providers or those providers with chronic medical conditions. Once a patient arrives emergently to the emergency department (ED) setting, ED providers must act promptly to evaluate these individuals for COVID-19 infection risk factors such as exposure, symptoms, and chronic medical conditions. However, some medical and surgical patients presenting emergently for evaluation are unable to provide a reliable medical history due to age, drugs, the absence of a next of kin, or altered mental status. Acutely traumatized patients often undergo computed tomography of the chest during their comprehensive evaluation. Adding a rapid bedside ultrasound of the chest as a research procedure could allow validation of ultrasound to help stratify medical and surgical patients into high and low risk of COVID-19 categories, with no radiation exposure, and far faster than current COVID-19 diagnostic PCR testing.

Aims: The project proposes to collect data that will inform a novel strategy to mitigate risk to providers by providing early, objective, and rapidly collected end organ data which will permit the stratification of pediatric trauma patients into low or high risk COVID-19 categories. The project will collect and evaluate lung ultrasound (US) findings in an expanded Focused Assessment with Sonography in Trauma (FAST) evaluation of the chest of pediatric trauma patients. The term "FAST+" is used to denote the use of FAST expanded to image the select lung fields in traumatized patients. The researchers hypothesize that FAST+ will result in identification of pulmonary findings indicative of COVID-19 infections and will significantly correlate with the gold standard derived from computed tomography (CT) performed in parallel in these traumatically injured patients.

ELIGIBILITY:
Inclusions:

1. Trauma patients presenting to our institution as trauma activation
2. Trauma patients presenting to our institution as trauma alerts

Exclusions:

1. Patients who require prompt surgical exploration based on physical exam findings (minimize delays in transport to the operating room)
2. Patients with an open chest injury

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All trauma patients evaluated at our institution that present as a trauma activation or alerts will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation of FAST+ pulmonary findings with active COVID infection | 12 months
  Will correlate FAST+ pulmonary findings and published CT findings noted in active COVID infection to determine if FAST+ is a suitable diagnostic tool in detecting active COVID infection. Plan to use FAST+ imaging findings to stratify patients into low or high-risk COVID-19 infection groups.

SECONDARY OUTCOMES:
Description of additional ancillary findings of the FAST+ examination among infected and non-infected patients | 12 months
  Exploratory outcomes will focus on description of additional ancillary findings of the FAST+ examination in those patients who later are determined to be COVID-19 positive compared to those determined to be COVID-19 negative (e.g., patterns of pleural space disease).

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Diaz-Miron, MD, Principal Investigator — University of Colorado/Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No